CLINICAL TRIAL: NCT01846806
Title: The Role of Bacterial Overgrowth and Delayed Intestinal Transit in Hepatic Encephalopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at NYUMC
Sponsor: NYU Langone Health (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-00570
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rifaximin (Experimental): Participants in Phase B will be administered 550 mg of Rifaximin two times a day for 14 days.
  Interventions: Other: Rifaximin

INTERVENTIONS:
Other: Rifaximin — Participants in Phase B will be administered 550 mg of Rifaximin two times a day for 14 days.

SUMMARY:
This is a prospective study designed to examine the role of bacterial overgrowth and delayed intestinal transit and the effect of Rifaximin with hepatic encephalopathy (HE). This study is divided into Phase A and Phase B. The purpose of Phase A is to test patients with cirrhosis to determine if they have bacterial overgrowth which may lead to slow intestinal transit and hepatic encephalopathy. The purpose of Phase B is to investigate whether the improvement found in patients with hepatic encephalopathy taking Rifaximin is also related to decreased bacterial overgrowth.

Subjects' mental capacity will be assessed at each visit via interview, brief mental status, questionnaires and psychometric evaluation. Any subject who appears to have lost capacity to continue participation, as evidenced by HE grade 2 or higher, a lack of attentiveness, concentration, or understanding of evaluation, will be discontinued from the study. Female subjects of childbearing potential will be asked to comply with the use of contraception during the Phase B study period as well as throughout the time they remain on study drug.

DETAILED DESCRIPTION:
This is a prospective study designed to examine the role of bacterial overgrowth and delayed intestinal transit and the effect of Rifaximin with hepatic encephalopathy (HE). This study is divided into Phase A and Phase B. The purpose of Phase A is to test patients with cirrhosis to determine if they have bacterial overgrowth which may lead to slow intestinal transit and hepatic encephalopathy. The purpose of Phase B is to investigate whether the improvement found in patients with hepatic encephalopathy taking Rifaximin is also related to decreased bacterial overgrowth. The target population is patients with chronic liver cirrhosis with or without symptoms of HE. Many patients may present with advanced cirrhosis and may be on the liver transplant list.

During Phase A, 20 patients will be asked to sign the informed consent form and will be assigned a subject number. They will be asked to provide demographic information, medical history, history of hospitalizations for HE, and HE medication use. They will undergo a complete physical examination, urine pregnancy test (women of childbearing potential), 12-lead EKG, grading of ascites, modified Child Pugh Score, MELD Score. They will also complete the following neuropsychological questionnaires: NCT, D-KEFS Trail Making Test, California Verbal Learning Test, WAIS-III Digit Symbol-Coding and Block Design, D-KEFS Stroop Color-Word Test, Evaluation of Constructional Apraxia, , and asterixis. During the evaluation visit (a minimum of 3 days after the Screening Visit) the following procedures will be performed: lab tests (chemistry and hematology panels). They will also complete the following questionnaires: Liver Disease Quality of Life Questionnaire, Fisk Fatigue Impact Score, Flatulence Survey, Epworth Sleepiness Scale. Finally, they will undergo a Lactulose Hydrogen Breath Test: This test is designed to evaluate both intestinal transit and bacterial overgrowth.

Participants in Phase B will be administered of 550 mg of Rifaximin two times a day for 14 days. Patients will be scheduled to come in on day 14 of the active study period. The follow up visit is day 28, where some of the tests described above will be repeated. During Phase B, patients will be asked to undergo a complete physical examination, a Neurological Examination [including calculation of modified Child Pugh and MELD Score NCT, and Trail Making Test], evaluation of constructional apraxia and asterixis. In addition, the researchers will make sure the patient meets eligibility criteria for participation in open label trial of Rifaximin. They will be administered the first dose study drug (Rifaximin) by study coordinator or investigator and they will be dispensed the study drug needed for the remainder of the trial and a diary for them to record daily flatulence. A urine pregnancy test will be performed within 48 hours of first study dose (for women of childbearing potential). During Day 14 and Day 28 visits, patients will have 1 tablespoon of blood drawn for measurement of the ammonia level and to monitor for potential blood clots. They will complete the NCT, Trails Test, Digit Symbol-Coding, Block Design, and Stroop Tests. They will also complete the Liver Disease Quality of Life Questionnaire, Fisk Fatigue Impact Score, Flatulence Survey (A diary will be provided to the patient with instructions on how to record flatulence experiences on a daily basis), and the Epworth Sleepiness Scale questionnaires. In addition, on Day 14, they will undergo another Lactulose Hydrogen Breath Test.

Subjects' mental capacity will be assessed at each visit via interview, brief mental status, questionnaires and psychometric evaluation. Any subject who appears to have lost capacity to continue participation, as evidenced by HE grade 2 or higher, a lack of attentiveness, concentration, or understanding of evaluation, will be discontinued from the study. Female subjects of childbearing potential will be asked to comply with the use of contraception during the Phase B study period as well as throughout the time they remain on study drug.

Following completion of the study, patients will be categorized by the degree of HE. To determine whether impaired intestinal transit and bacterial overgrowth are associated with severity of HE, multivariate analysis will be performed to determine whether the independent factors of liver disease severity, intestinal transit, and bacterial overgrowth are significant predictors of the presence and severity of HE. Also, to determine whether treatment with Rifaximin improves bacterial overgrowth, ammonia levels, and HE, changes in Breath Test analysis be correlated will be correlated with changes in ammonia levels and HE.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients with HCV cirrhosis will be screened for participation in the study
* Ability to complete Number Connection Test
* Creatinine <1.5mg/dL
* Able to provide informed consent
* Patients determined to possibly meet the West Haven criteria grade 0 or 1 for HE

Exclusion Criteria:

* Active interferon therapy
* History of alcohol abuse within six months
* Active gastrointestinal bleeding
* Use of agents that alter intestinal motility, e.g., methadone, cholestyramine, Tricyclic antidepressants, etc.
* Use of Neomycin or other antibiotics within the past 2 weeks
* Pregnancy
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Lactulose Hydrogen Breath Test | Day 3 and Day 14
  This test is designed to evaluate both intestinal transit and bacterial overgrowth. Subjects will be asked to breathe into a collection bag, drink 10g of lactulose that has been mixed with 8 oz of water, breathe again into the collection bag after waiting 20 minutes and then again every 10 minutes for a total of 2 hours.

SECONDARY OUTCOMES:
Hepatic Encephalopathy | Phase A (Screening), Phase B (Day 1, Day 14, and Day 28)
  Subjects will be administered the Number Connection Test, WAIS-III Block Design and Digit Symbol Coding, DKEFS Trail Making and Color Word Interference, and California Verbal Learning Test-II
Quality of Life | Phase A (Evaluation), Phase B (Day 1, Day 14, and Day 28)
  Subjects will be asked to complete the Beck Depression Inventory-II, Liver Disease Quality of Life Questionnaire, Fisk Fatigue Impact Scale, Epworth Sleepiness Scale, and Hamilton Depression Inventory
Laboratory Tests | 3 days
  Results will be evaluated for the following lab tests: blood chemistry (including ammonia and other potential toxins) and hematology panels

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Medical Center, New York, New York, United States